CLINICAL TRIAL: NCT04153487
Title: Role of Ascorbic Acid Infusion in Critically Ill Patients With Transfusion Related Acute Lung Injury
Acronym: ASTRALI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASTRALI
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2021-05

CONDITIONS: Acute Lung Injury, Transfusion Related
Keywords: Transfusion Reaction; Transfusion Related Complication; Acute Lung Injury; Critical Care
MeSH Terms: conditions — Transfusion-Related Acute Lung Injury; Transfusion Reaction; Acute Lung Injury | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASTRALI Group (Experimental): ASTRALI (AScorbic acid in TRALI) group (n=40)
  Interventions: Drug: Ascorbic Acid Injectable Product
- Control Group (Placebo Comparator): Control group (n=40)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic Acid Injectable Product — Intermittent Intravenous Infusion of Ascorbic Acid (Vitamin C) 2.5 gm / 6 hours for 96 hours
  Other Names: Vitamin C
  Arms: ASTRALI Group
Drug: Placebo — Placebo saline / 6 hours for 96 hours
  Other Names: Normal saline
  Arms: Control Group

SUMMARY:
TRALI was defined as "acute noncardiogenic pulmonary edema typically occurs ≤ 6 hours following transfusion of plasma-containing blood products, such as packed red blood cells, fresh frozen plasma, platelets, or cryoprecipitate." In critically ill patients, TRALI remains the leading cause of transfusion-related fatalities and is accompanied by a very significant morbidity and mortality. Survival in such patients is as low as 53% compared with 83% in acute lung injury (ALI) controls.

The incidence of TRALi is likely underreported. In densely populated developing countries, incidence has not decreased due to lack of male-only strategy for plasma donation.

TRALI is associated with systemic inflammation characterized by low anti-inflammatory cytokine as interleukin (IL)-10, increased pro-inflammatory cytokine as IL-8. Regulation of inflammation should include avoidance of overproduction of inflammatory mediators. So, it can be dampened not only by increasing IL-10 but also by decreasing IL-1β release. C-reactive protein (CRP) is an acute phase protein which is up-regulated during infections and inflammation. CRP was recently identified as a novel first hit in TRALI.

Till now, there is no established treatment for TRALI beyond supportive care and monitoring. Recently, potential therapies have been reviewed, and it was concluded that the most promising therapeutic strategies are IL-10 therapy, downregulation of CRP levels, targeting reactive oxygen species (ROS) or blocking IL-8 receptors. So, antioxidants (such as high dose vitamins), were recommended for future studies as potentially effective treatment.

Vitamin C hypovitaminosis is observed in 70% of critically ill despite receiving recommended daily doses.

The aim of this study is to investigate the role of intravenous vitamin C (ascorbic acid) as a targeted therapy for transfusion related acute lung injury (TRALI) in critically ill patients in terms of IL-8, IL-10, CRP, SOD, malondialdehyde (MDA), vasopressor use, duration of mechanical ventilation, ICU length of stay, 7-days mortality and 28-days mortality.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. The minimum required sample size is estimated to be 40 patients for each group.
3. Full written informed consent will be taken from all patients or their next of kin to participate in this study.
4. All patients will be subjected directly at time of enrollment to the following;

   * Complete history taking and demographic data
   * The potential recipient risk factors for TRALI.
   * The initial cause of ICU admission and the blood products received.
   * Complete physical examination including chest auscultations.
   * Vital signs
   * Routine laboratory investigations
   * Brain natriuretic peptide level
   * Troponin T
   * Hypoxic index
   * Acute Physiology and Chronic Health Evaluation version II (APACHE II) score.
   * Sequential Organ Failure Assessment (SOFA) score.
   * Kidney Disease Improving Global Outcomes (KDIGO) criteria.
   * Child Pugh score.
   * Chest radiography and transthoracic echocardiography.
5. Samples will be drawn to measure the initial values of ascorbate level, plasma IL-8, IL-10, IL-1β, SOD, MDA and serum CRP.
6. Eighty patients with confirmed TRALI (n=80) will be enrolled from critical care units (tertiary hospitals). Then, in addition to their supportive and standard care, they will be randomized (computer sheet) into two groups:

   * ASTRALI (AScorbic acid in TRALI) group (n=40) will receive 2.5 gm vitamin C intravenously every 6 hrs for 96 hrs from diagnosis.
   * Control group (n=40) will receive placebo in similar regimen.
7. All patients will be followed up and treated during the study time. All relevant routine investigations, supportive measures, medications and ventilatory data will be recorded.
8. All possible adverse events will be monitored, recorded and managed directly. Hyperoxaluria, microscopic calcium-oxalate crystallization or oxalate nephropathy will be monitored, recorded and managed directly.
9. After 96 hrs, resampling for ascorbate level and the same biomarkers will be done.
10. Measuring the study secondary outcomes will include vasopressor use, duration of mechanical ventilation, ICU length of stay, 7-days mortality and 28-days mortality.
11. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 - 64 years) critically ill patients diagnosed with transfusion related acute lung injury (TRALI), at the time of enrollment or maximum 6 hours before, according to the National Heart, Lung and Blood Institute (NHLBI) Working Group definitions and or the Canadian Consensus Conference criteria (29, 30) as the following criteria;

  * No evidence of ALI prior to transfusion.
  * Onset of ALI ≤ 6 hours following cessation of transfusion.
  * Hypoxemia, defined as the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) ≤ 300 mmHg or oxygen saturation ≤ 90% on room air.
  * Radiographic evidence of bilateral infiltrates.
  * No evidence of left atrial hypertension.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Hypernatremia or known hypersensitivity to the study drug.
* Parenteral nutrition (total/partial) containing vitamin C.
* Active renal stone or history of urolithiasis.
* Acute Kidney Injury.
* Glucose 6 phosphate dehydrogenase deficiency, iron and copper storage diseases.
* Immunocompromised patients (cancer or patients on immunosuppressive drugs).
* Moribund patient not expected to survive 24 hours .
* Home mechanical ventilation (via tracheotomy or noninvasive) except for Continuous Positive Airway Pressure/ Bilevel Positive Airway Pressure (CPAP/BIPAP) used only for sleep-disordered breathing .

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Interleukin-8 (IL-8) | 96 hrs
  Plasma level of IL-8
Interleukin-10 (IL-10) | 96 hrs
  Plasma Level of IL-10
C-reactive protein (CRP) | 96 hrs
  Serum level of CRP
Superoxide Dismutase (SOD) | 96 hrs
  Plasma Level of SOD
Malondialdehyde (MDA) | 96 hrs
  Plasma level of MDA

SECONDARY OUTCOMES:
Vasopressor use (days) | up to 28 days
  Duration of circulatory support
Duration of Mechanical Ventilation (days) | up to 28 days
  Duration of ventilatory support
ICU length of stay (days) | Up to 28 days
  Length of stay in ICU
7-days Mortality | 7 days
  All cause mortality
28-days Mortality | 28 days
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Gamal A Omran, PHD, Study Director — Professor of Biochemistry, Damanhour University.; Mohamed M Megahed, MD, Study Director — Professor of Critical Care Medicine, Alexandria University.; Tamer N Zakhary, MD, Study Chair — Ass. Professor of Critical Care Medicine, Alexandria University.; Amira B Kassem, PHD, Study Chair — Lecturer of Clinical Pharmacy, Damanhour University.; Islam E Ahmed, PharmD, Principal Investigator — Clinical Pharmacy Specialist, Damanhour University.
Locations (1):
- Damanhour University, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No
The summary of all relevant data

REFERENCES:
- [Background] Peters AL, Van Stein D, Vlaar AP. Antibody-mediated transfusion-related acute lung injury; from discovery to prevention. Br J Haematol. 2015 Sep;170(5):597-614. doi: 10.1111/bjh.13459. Epub 2015 Apr 28. PMID 25921271
- [Background] Vlaar AP, Juffermans NP. Transfusion-related acute lung injury: a clinical review. Lancet. 2013 Sep 14;382(9896):984-94. doi: 10.1016/S0140-6736(12)62197-7. Epub 2013 May 1. PMID 23642914
- [Background] Roubinian N. TACO and TRALI: biology, risk factors, and prevention strategies. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):585-594. doi: 10.1182/asheducation-2018.1.585. Epub 2018 Dec 14. PMID 30570487
- [Background] Peters AL, van Hezel ME, Juffermans NP, Vlaar AP. Pathogenesis of non-antibody mediated transfusion-related acute lung injury from bench to bedside. Blood Rev. 2015 Jan;29(1):51-61. doi: 10.1016/j.blre.2014.09.007. Epub 2014 Sep 20. PMID 25277811
- [Background] Andreu G, Boudjedir K, Muller JY, Pouchol E, Ozier Y, Fevre G, Gautreau C, Quaranta JF, Drouet C, Rieux C, Mertes PM, Clavier B, Carlier M, Sandid I. Analysis of Transfusion-Related Acute Lung Injury and Possible Transfusion-Related Acute Lung Injury Reported to the French Hemovigilance Network From 2007 to 2013. Transfus Med Rev. 2018 Jan;32(1):16-27. doi: 10.1016/j.tmrv.2017.07.001. Epub 2017 Jul 15. PMID 28864336
- [Background] Vlaar AP, Binnekade JM, Prins D, van Stein D, Hofstra JJ, Schultz MJ, Juffermans NP. Risk factors and outcome of transfusion-related acute lung injury in the critically ill: a nested case-control study. Crit Care Med. 2010 Mar;38(3):771-8. doi: 10.1097/CCM.0b013e3181cc4d4b. PMID 20035217
- [Background] Vlaar APJ, Toy P, Fung M, Looney MR, Juffermans NP, Bux J, Bolton-Maggs P, Peters AL, Silliman CC, Kor DJ, Kleinman S. An update of the transfusion-related acute lung injury (TRALI) definition. Transfus Clin Biol. 2019 Nov;26(4):354-356. doi: 10.1016/j.tracli.2019.05.007. Epub 2019 Jun 12. No abstract available. PMID 31221537
- [Background] Toy P, Gajic O, Bacchetti P, Looney MR, Gropper MA, Hubmayr R, Lowell CA, Norris PJ, Murphy EL, Weiskopf RB, Wilson G, Koenigsberg M, Lee D, Schuller R, Wu P, Grimes B, Gandhi MJ, Winters JL, Mair D, Hirschler N, Sanchez Rosen R, Matthay MA; TRALI Study Group. Transfusion-related acute lung injury: incidence and risk factors. Blood. 2012 Feb 16;119(7):1757-67. doi: 10.1182/blood-2011-08-370932. Epub 2011 Nov 23. PMID 22117051
- [Background] Semple JW, Rebetz J, Kapur R. Transfusion-associated circulatory overload and transfusion-related acute lung injury. Blood. 2019 Apr 25;133(17):1840-1853. doi: 10.1182/blood-2018-10-860809. Epub 2019 Feb 26. PMID 30808638
- [Background] Roubinian NH, Looney MR, Kor DJ, Lowell CA, Gajic O, Hubmayr RD, Gropper MA, Koenigsberg M, Wilson GA, Matthay MA, Toy P, Murphy EL; TRALI Study Group. Cytokines and clinical predictors in distinguishing pulmonary transfusion reactions. Transfusion. 2015 Aug;55(8):1838-46. doi: 10.1111/trf.13021. Epub 2015 Feb 23. PMID 25702590
- [Background] Semple JW, McVey MJ, Kim M, Rebetz J, Kuebler WM, Kapur R. Targeting Transfusion-Related Acute Lung Injury: The Journey From Basic Science to Novel Therapies. Crit Care Med. 2018 May;46(5):e452-e458. doi: 10.1097/CCM.0000000000002989. PMID 29384784
- [Background] Ducharme-Crevier L, Lacroix J. Interleukin-1 Receptor Antagonist and Interleukin-1beta: Risk Marker or Risk Factor for Pediatric Acute Respiratory Distress Syndrome? Pediatr Crit Care Med. 2018 Oct;19(10):993-995. doi: 10.1097/PCC.0000000000001713. No abstract available. PMID 30281566
- [Background] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Background] Kapur R, Kim M, Shanmugabhavananthan S, Liu J, Li Y, Semple JW. C-reactive protein enhances murine antibody-mediated transfusion-related acute lung injury. Blood. 2015 Dec 17;126(25):2747-51. doi: 10.1182/blood-2015-09-672592. Epub 2015 Oct 9. PMID 26453659
- [Background] Kapur R, Kim M, Rondina MT, Porcelijn L, Semple JW. Elevation of C-reactive protein levels in patients with transfusion-related acute lung injury. Oncotarget. 2016 Nov 22;7(47):78048-78054. doi: 10.18632/oncotarget.12872. PMID 27793007
- [Background] McNamara R, Deane AM, Anstey J, Bellomo R. Understanding the rationale for parenteral ascorbate (vitamin C) during an acute inflammatory reaction: a biochemical perspective. Crit Care Resusc. 2018 Sep;20(3):174-179. No abstract available. PMID 30153778
- [Background] Carr AC, Rosengrave PC, Bayer S, Chambers S, Mehrtens J, Shaw GM. Hypovitaminosis C and vitamin C deficiency in critically ill patients despite recommended enteral and parenteral intakes. Crit Care. 2017 Dec 11;21(1):300. doi: 10.1186/s13054-017-1891-y. PMID 29228951
- [Background] Margaritelis NV, Paschalis V, Theodorou AA, Vassiliou V, Kyparos A, Nikolaidis MG. Rapid decreases of key antioxidant molecules in critically ill patients: A personalized approach. Clin Nutr. 2020 Apr;39(4):1146-1154. doi: 10.1016/j.clnu.2019.04.029. Epub 2019 Apr 29. PMID 31080038
- [Background] Carr AC, Maggini S. Vitamin C and Immune Function. Nutrients. 2017 Nov 3;9(11):1211. doi: 10.3390/nu9111211. PMID 29099763
- [Background] Hartmann SE, Waltz X, Kissel CK, Szabo L, Walker BL, Leigh R, Anderson TJ, Poulin MJ. Cerebrovascular and ventilatory responses to acute isocapnic hypoxia in healthy aging and lung disease: effect of vitamin C. J Appl Physiol (1985). 2015 Aug 15;119(4):363-73. doi: 10.1152/japplphysiol.00389.2015. Epub 2015 Jun 18. PMID 26089546
- [Background] Reynolds PS, Fisher BJ, McCarter J, Sweeney C, Martin EJ, Middleton P, Ellenberg M, Fowler E, Brophy DF, Fowler AA 3rd, Spiess BD, Natarajan R. Interventional vitamin C: A strategy for attenuation of coagulopathy and inflammation in a swine multiple injuries model. J Trauma Acute Care Surg. 2018 Jul;85(1S Suppl 2):S57-S67. doi: 10.1097/TA.0000000000001844. PMID 29538225
- [Background] Wang Y, Lin H, Lin BW, Lin JD. Effects of different ascorbic acid doses on the mortality of critically ill patients: a meta-analysis. Ann Intensive Care. 2019 May 20;9(1):58. doi: 10.1186/s13613-019-0532-9. PMID 31111241
- [Background] Rozemeijer S, Spoelstra-de Man AME, Coenen S, Smit B, Elbers PWG, de Grooth HJ, Girbes ARJ, Oudemans-van Straaten HM. Estimating Vitamin C Status in Critically Ill Patients with a Novel Point-of-Care Oxidation-Reduction Potential Measurement. Nutrients. 2019 May 8;11(5):1031. doi: 10.3390/nu11051031. PMID 31071996
- [Background] Buehner M, Pamplin J, Studer L, Hughes RL, King BT, Graybill JC, Chung KK. Oxalate Nephropathy After Continuous Infusion of High-Dose Vitamin C as an Adjunct to Burn Resuscitation. J Burn Care Res. 2016 Jul-Aug;37(4):e374-9. doi: 10.1097/BCR.0000000000000233. PMID 25812044
- [Background] Schorah CJ, Downing C, Piripitsi A, Gallivan L, Al-Hazaa AH, Sanderson MJ, Bodenham A. Total vitamin C, ascorbic acid, and dehydroascorbic acid concentrations in plasma of critically ill patients. Am J Clin Nutr. 1996 May;63(5):760-5. doi: 10.1093/ajcn/63.5.760. PMID 8615361
- [Background] Long CL, Maull KI, Krishnan RS, Laws HL, Geiger JW, Borghesi L, Franks W, Lawson TC, Sauberlich HE. Ascorbic acid dynamics in the seriously ill and injured. J Surg Res. 2003 Feb;109(2):144-8. doi: 10.1016/s0022-4804(02)00083-5. PMID 12643856
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] de Grooth HJ, Manubulu-Choo WP, Zandvliet AS, Spoelstra-de Man AME, Girbes AR, Swart EL, Oudemans-van Straaten HM. Vitamin C Pharmacokinetics in Critically Ill Patients: A Randomized Trial of Four IV Regimens. Chest. 2018 Jun;153(6):1368-1377. doi: 10.1016/j.chest.2018.02.025. Epub 2018 Mar 6. PMID 29522710
- [Background] Toy P, Popovsky MA, Abraham E, Ambruso DR, Holness LG, Kopko PM, McFarland JG, Nathens AB, Silliman CC, Stroncek D; National Heart, Lung and Blood Institute Working Group on TRALI. Transfusion-related acute lung injury: definition and review. Crit Care Med. 2005 Apr;33(4):721-6. doi: 10.1097/01.ccm.0000159849.94750.51. PMID 15818095
- [Background] Kleinman S, Caulfield T, Chan P, Davenport R, McFarland J, McPhedran S, Meade M, Morrison D, Pinsent T, Robillard P, Slinger P. Toward an understanding of transfusion-related acute lung injury: statement of a consensus panel. Transfusion. 2004 Dec;44(12):1774-89. doi: 10.1111/j.0041-1132.2004.04347.x. No abstract available. PMID 15584994
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637
- [Background] Wagner DP, Draper EA. Acute physiology and chronic health evaluation (APACHE II) and Medicare reimbursement. Health Care Financ Rev. 1984;Suppl(Suppl):91-105. PMID 10311080
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Kdigo AJKIS. Work Group. KDIGO clinical practice guideline for acute kidney injury. 2012;2(1):1-138.
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913
- [Background] Klimant E, Wright H, Rubin D, Seely D, Markman M. Intravenous vitamin C in the supportive care of cancer patients: a review and rational approach. Curr Oncol. 2018 Apr;25(2):139-148. doi: 10.3747/co.25.3790. Epub 2018 Apr 30. PMID 29719430
- [Derived] Kassem AB, Ahmed I, Omran G, Megahed M, Habib T. Role of ascorbic acid infusion in critically ill patients with transfusion-related acute lung injury. Br J Clin Pharmacol. 2022 May;88(5):2327-2339. doi: 10.1111/bcp.15167. Epub 2022 Jan 7. PMID 34866234